CLINICAL TRIAL: NCT06651385
Title: Pilot of Exercise and Asthma Control
Acronym: PEAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Kate M Huether, Principal Investigator, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002796
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Asthma; Obesity
Keywords: Exercise
MeSH Terms: conditions — Asthma; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Remote digital therapeutic exercise program (Experimental)
  Interventions: Other: Remote digital therapeutic exercise program

INTERVENTIONS:
Other: Remote digital therapeutic exercise program — Participants will be introduced to the digital therapeutic exercise program during Screening and Consent (Visit 0, V0). Participants will be provided with an orientation to the Vitala platform and assistance will be offered in the download and access to the application, as needed. The study team will ensure access has been obtained via the health care professionals' dashboard on the Vitala app. Information obtained in the assessments outlined above will inform the tailored exercise prescription to meet the participant's needs. Participants will be encouraged to complete a total of 150 minutes of remote exercise sessions each week for 12 weeks via the Vitala platform. Participants will receive daily notifications to remind them to complete their assigned daily exercises.

SUMMARY:
This will be a pilot, single arm, un-blinded study of a remote digital therapeutic exercise program in adults with obesity and poorly controlled asthma. Participants will be recruited from the University of Vermont Medical Center adult Pulmonary Clinic, Internal Medicine Clinic, and from the greater community via flyers and referrals, as needed. The primary outcome of interest will be the feasibility and acceptability of a remote digital therapeutic exercise program using a mobile application, called Vitala. Vitala is a FDA Registered, HIPAA Compliant CE-marked MDR class 1 medical device developed by doctors and physiotherapists. It is a mobile application tool that enables health care providers to prescribe and monitor diagnosis-specific exercise prescriptions that allows patients to remotely access their tailored therapeutic exercise program. URL: Medical exercise and digital rehabilitation - Vitala

Feasibility and acceptability will be defined as ≥60% of subjects enrolled in the exercise program completing, on average, ≥50% (≥75 minutes/ week) of the digital exercise program during their 12-week period, respectively. The secondary outcome of interest will be the efficacy of a remote digital therapeutic exercise program in participants with obesity and poorly controlled asthma by comparing asthma symptoms before, during, and at the end of the intervention. Efficacy will be defined as ≥30% of subjects who achieving a minimal clinically important difference in Asthma Control Test scores (defined as increase of ≥3 points[31]).

The Investigators plan to enroll participants on a rolling basis. Prospective participants will be contacted by phone, mail, or e-mail to establish interest and eligibility in the study. Once confirmed interested and eligible to participate in the study, they will be scheduled for eConsent and enrollment in the study (V0). Participants will receive a tailored exercise prescription unique to their individual needs, space, and available equipment and will be encouraged to complete 150 minutes of activity per week via their customized exercise program through the Vitala platform remotely for 12 weeks. Participants will be contacted when the program has been made available to them for program start, which will also be guided based on the participant's availability and preferred program start date (P0). During the 12 week exercise program, participants will have 3 remote contacts/visits (RC, V1, and 2), approximately every 4 - 6 weeks, over the 12 week intervention period including a final remote visit (V2) after completion of the program to assess adherence to the program, asthma control, and asthma-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of asthma on regular prescribed controller therapy for 3 months prior to enrollment (per EMR or self-report)
* Age: ≥18 years of age
* Obese: BMI ≥30 kg/m2
* Poorly controlled asthma (defined as one or more of the following criteria:
* Asthma Control Test Score ≤19, or
* Use of rescue inhaler on average >2 uses/week for preceding month, or
* Nocturnal asthma awakening on average ≥1 times/week in preceding month, or
* ED/hospital visit or prednisone course for asthma in past six months
* Ability and willingness to provide informed consent
* Internet access on a mobile smart phone to access the digital exercise program

Exclusion Criteria:

* Any condition that precludes participation in regular exercise as judged by the investigator and/or study physician
* Pregnancy (by self-report)
* Active participation in another exercise or weight loss program, or within 30 days prior to enrollment
* Current use of prescription weight loss medication, or within 30 days or 5- half lives, whichever is longer, prior to enrollment.
* Failing to meet criteria on the PAR-Q+ screening questionnaire for safe exercise [32, 33]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the feasibility and acceptability of a remote digital therapeutic exercise program in people with obesity and poorly controlled asthma. | 12 weeks
  Successful feasibility will be defined as ≥60% of subjects enrolled in the exercise program completing, on average, ≥50% (≥75 minutes/ week) of the digital exercise program during their 12-week period.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study to examine the feasibility of an exercise program in subjects with poorly controlled asthma and obesity. The data may be used for future research by the local study team only for projects examining the impact of exercise on asthma control.